CLINICAL TRIAL: NCT04010825
Title: Impact of Hypnosis Intervention Focused on the Emotional Dimension of Dyspnea on the Maintenance of Benefits for Patients With COPD After a Pulmonary Rehabilitation: A Multicenter Randomized Controlled Clinical Study
Brief Title: Impact of Hypnosis Intervention on the Emotional Dimension of Dyspnea in Patients With COPD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DYSPNEMO
Record Dates: First submitted 2019-06-26; First posted 2019-07-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Dyspnea; Pulmonary rehabilitation; Physical activity; Hypnosis; Anxiety; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Arm (Experimental): In parallel with an inpatient pulmonary rehabilitation program, nine visits will be carried out :
  * V0 : an inclusion visit
  * V1 : a randomization visit
  * V2 to V6 : five visits with hypnosis sessions
  * V7 : a end-stay visit
  * V8 : a 6-month post-rehabilitation visit ( by phone call)
  The five hypnosis sessions (V2 to V6) will be spread over three weeks of rehabilitation program (1 to 2 hypnosis sessions per week).
  For V1, V7 and V8 : questionnaires will be filled about : quality of life (CAT questionnaire), the three dimensions of dyspnea (mMRC, LCADL and MDP questionnaires), anxiety and depression (HADS questionnaire), post-traumatic stress ( PCLS questionnaire), sedentarity and physical activity (SIMPAQ questionnaire). Other data will be also collected on : previous experiences with hypnosis, self-hypnosis and relaxation, number of exacerbations and hospitalizations in the past 6 months, drug treatment, psychotropic drug use and dosage and psychological follow-up.
  Interventions: Other: Hypnosis intervention focused on the emotional dimension of the dyspnea
- Control Arm (No Intervention): In parallel with an inpatient pulmonary rehabilitation program, no additional intervention will be carry out and four visits will be carried out :
  * V0 : an inclusion visit
  * V1 : a randomization visit
  * V7 : a end-stay visit
  * V8 : a 6-month post-rehabilitation visit ( by phone call)
  For V1, V7 and V8 : questionnaires will be filled about : quality of life (CAT questionnaire), the three dimensions of dyspnea (mMRC, LCADL and MDP questionnaires), anxiety and depression (HADS questionnaire), post-traumatic stress ( PCLS questionnaire), sedentarity and physical activity (SIMPAQ questionnaire). Other data will be also collected on : previous experiences with hypnosis, self-hypnosis and relaxation, number of exacerbations and hospitalizations in the past 6 months, drug treatment, psychotropic drug use and dosage and psychological follow-up.

INTERVENTIONS:
Other: Hypnosis intervention focused on the emotional dimension of the dyspnea — Individual hypnosis sessions will be for 1 hour. Each hypnosis session will be standardized and evaluated using a script and an observation grid ( Visual Analogic Scale comfort, patient's hypnotic state...) written in collaboration with experts from Institut Milton Hyland Erickson Toulouse France (IMHETO).
  Arms: Hypnosis Arm

SUMMARY:
The purpose of the clinical study is to compare the effect of hypnosis intervention on the emotional dimension of the dyspnea during a pulmonary rehabilitation program to the pulmonary rehabilitation program alone. This study will determine if the hypnosis intervention will lead to better maintenance of benefits obtained than the original described method.

DETAILED DESCRIPTION:
While physical activity level is the best predictor of life expectancy for patients with chronic obstructive pulmonary disease (COPD), the majority of patients have physical activity levels well below guidelines. One of the main barriers to regular activity is anxiety related to dyspnea. Defined as a subjective experience of discomfort during breathing, dyspnea is described as a multidimensional phenomenon integrating both the impact dimension (daily disability), the sensory dimension (intensity of dyspnea) and the emotional dimension (unpleasant and anxiety-aspects). The most effective treatment to reduce dyspnea is pulmonary rehabilitation. An overall improvement in dyspnea, and more specifically in its emotional dimension, has been achieved by reducing dyspnea anxiety. By reducing one of the major barriers to regular physical activity, the level of post-rehabilitation physical activity should also be improved. However, paradoxically, many studies have reported that there has been no change in the level of physical activity of patients in post-rehabilitation. A possible hypothesis to explain this decoupling between the improvement of the emotional dimension of dyspnea and the absence of behavioral modification, lies in the disappearance of the effects once at home. Indeed, during a pulmonary rehabilitation stay, patients practice under health professionals' supervision and advices with regular feedback on their abilities. When patients return home left on their own again, dyspnea anxiety is likely to reappear and motivation may not be enough.

Several techniques have been proposed to complement traditional interventions in order to strengthen rehabilitation effects. Unfortunately, these are not effective. The use of hypnosis as a complement to rehabilitation programs is a promising perspective to maintain the benefits on the emotional dimension of dyspnea after a rehabilitation program. Its benefits have already been demonstrated in the reduction of acute and chronic pains, in a long-term effectiveness using self-hypnosis techniques. These ensure the continuity of remote management of the intervention. Given the analogy between pain and dyspnea, hypnosis could therefore constitute a therapeutic solution as a complement to rehabilitation to durably reduce dyspnea anxiety in patients with COPD, and promote a better behavior at middle and long term.

The investigators hypothesize that hypnosis used in addition to a 4-week pulmonary rehabilitation program will maintain the benefits on the emotional dimension of dyspnea at 6 months in the experimental group compared to a control group.

The main objective is to evaluate the impact of a hypnosis intervention during a pulmonary rehabilitation program on the emotional dimension of dyspnea 6 months after patients return home (T2).

ELIGIBILITY:
Inclusion Criteria:

* Admitted for a 4-week inpatient pulmonary rehabilitation program
* COPD diagnosis with a value of the first second of forced expiration (FEV1) < 80% of theoretical values
* 40 and 75 years old
* Reading and writing skills

Exclusion Criteria:

* Inability to answer a questionnaire
* Patient with psychosis or psychiatric disorders with delusions (or delusions history)
* Pregnant women
* Protected adults
* Participation in another study, with the exception of observational studies

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Differential of the emotional dimension of dyspnea 6 months after pulmonary rehabilitation (PR) | Change from baseline (T0) to 6 month follow-up (T2)
  Assessing differential of the emotional dimension of dyspnea score on the Multidimensional Dyspnea Profile scale (MDP questionnaire Meek et al 2012) 6 months after pulmonary rehabilitation (PR).
  MDP is a 11 items questionnaire. Each item is graded 0-10. 5 items are devoted to the emotional dimension of dyspnea. High scores indicate high prevalence of symptoms.
  As proposed by Morélot-Panzini et al in 2016, for filling it up, patient will be asked to focus on his worst dyspnea experience that happened oin the last two weeks.

SECONDARY OUTCOMES:
Differential of the emotional dimension of dyspnea from baseline to PR end-stay and from PR end-stay to 6 months after PR | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) and from T1 to 6 month follow-up (T2)
  Assessing differential of the emotional dimension of dyspnea score on the Multidimensional Dyspnea Profile scale (MDP questionnaire Meek et al 2012) from baseline to PR end-stay and from PR end-stay to 6 months after PR .
  MDP is a 11 items questionnaire. Each item is graded 0-10. 5 items are devoted to the emotional dimension of dyspnea. High scores indicate high prevalence of symptoms.
  As proposed by Morélot-Panzini et al in 2016, for filling it up, patient will be asked to focus on his worst dyspnea experience that happened oin the last two weeks.
Differential of the impact dimension of dyspnea | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the impact dimension of dyspnea score on the modified Medical Research Council scale ( mMRC questionnaire) and on the London Chest of Activity Daily Living (LCADL) at the PR end-stay and 6 months after PR.
  mMRC is a 1 item questionnaire graded 0-4. High score indicates high prevalence of symptoms.
  LCADL is a15-item, self-administered questionnaire which allows an evaluation of dyspnea in patients with COPD during daily activities divided into four components: self-care, domestic, physical, and leisure. Patients could score from 0: "I would not do anyway" to 5: "I need someone else to do this". LCADL score is calculated by aggregating the points assigned to each question, with a higher score representing maximal disability.
Differential of the sensory dimension of dyspnea | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the sensory dimension of dyspnea score on the Multidimensional Dyspnea Profile scale (MDP questionnaire Meek et al 2012) at the PR end-stay and 6 months after PR.
  MDP is a 11 items questionnaire. Each item is graded 0-10. 6 items are devoted to the sensory dimension of dyspnea. High scores indicate high prevalence of symptoms.
  As proposed by Morélot-Panzini et al in 2016, for filling it up, patient will be asked to focus on his worst dyspnea experience that happened oin the last two weeks.
Differential of the post-traumatic stress disorder | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the post-traumatic stress disorder score (PCLS questionnaire) at the PR end-stay and 6 months after PR.
  PCLS is a 17 items questionnaire. Each item is graded 1-5. A score higher than 44 indicates patient has a post-traumatic disorder as defined by in Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV) (Weathers et al, 1993).
Differential of the quality of life | Changes from baseline (T0) to at the end of the 4-weeks PR , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the quality of life score (COPD Assessment Test-CAT questionnaire) at the PR end-stay and 6 months after PR.
  CAT is a COPD specific questionnaire including 8 items. Each item is graded 0-5. Global score is comprised between 0 and 40. Higher global score is higher COPD impact on patient's quality of life is.
Differential of the anxiety and depression | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the anxiety and depression score (Hospital Anxiety and Depression Scale -HADS questionnaire) at the PR end-stay and 6 months after PR.
  HADS is a 14 items questionnaire (7 items for anxiety and 7 items for depression). Each item is graded 0-3. A score higher than 7 indicates anxiety and/or depression
Differential of the physical activity and sedentarity levels | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  Assessing differential of the physical activity and sedentarity levels (Simple Physical Activity Questionnaire (SIMPAQ) at the PR end-stay and 6 months after PR.
  SIMPAQ is a 5 items questionnaire assessing in the last two weeks physical activity levels, sedentary times and time in bed.
Questionnaire for assessing psychotropic drug quantity and dosage | Changes from baseline (T0) to at the end of the 4-weeks PR (T1) , from T0 to 6 month follow-up (T2) and from T1 to 6 month follow-up (T2)
  A short questionnaire will be used for assessing differential of psychotropic drug quantity and dosage at the PR end-stay and 6 months after PR.
Number of exacerbations and hospitalizations | Changes from baseline (T0) to 6 month follow-up (T2)
  Assessing differential of number of exacerbations and hospitalizations 6 months after PR.
  Number of exacerbations and hospitalizations happened during the 6 last months will be indicated at T0 (baseline) and at T2 (6 month follow-up)
Hypnosis frequency | Changes from baseline (T0) to 6 month follow-up (T2)
  Assessing hypnosis frequency 6 months after PR.
Number of participants with previous hypnosis experiences | Months or/and years before PR baseline (T0)
  A questionnaire will be used for assessing patient's previous hypnosis experiences (previous to PR). (counting)
Self-Hypnosis frequency | Changes from baseline (T0) to 6 month follow-up (T2)
  Assessing self-hypnosis frequency 6 months after PR.
Number of participants with previous self-hypnosis experiences | Months or/and years before PR baseline (T0)
  A questionnaire will be used for assessing patient's previous self-hypnosis experiences (previous to PR). (counting)
Relaxation methods frequency | Changes from baseline (T0) to 6 month follow-up (T2)
  Assessing relaxation methods frequency 6 months after PR.
Number of participants with previous relaxation methods experiences | Months or/and years before PR baseline (T0)
  A questionnaire will be used for assessing patient's previous relaxation methods experiences (previous to PR). (counting)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Castanyer, Principal Investigator — 5 SANTE - Clinique du Souffle la Solane; Nelly Heraud, PhD, Study Director — 5 Santé
Locations (2):
- France (2):
  - Clinique du Souffle la Vallonie, Lodève
  - Clinique du Souffle la Solane, Osséja

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandes N, Alexandre F, Molinier V, Castanyer A, Moine E, Heraud N. Effect of dyspnoea-oriented hypnosis as an adjunct to pulmonary rehabilitation on the affective dimension of dyspnoea and physical activity level: a randomised controlled trial. ERJ Open Res. 2026 Feb 2;12(1):00621-2025. doi: 10.1183/23120541.00621-2025. eCollection 2026 Jan. PMID 41635580